CLINICAL TRIAL: NCT03394300
Title: Accuracy of Intraocular Lens Power in High Myopia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, salma safwat abdelhady mangora, ophthalmology resident, Assiut University
Other Study IDs: 29110202500209
Record Dates: First submitted 2017-12-29; First posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: High Myopia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: iol power calculation — iol power calculation in high myopia

SUMMARY:
evaluation of the accuracy of iol power in high myopia using different biometry formula & iol master

DETAILED DESCRIPTION:
High myopia or pathological myopia is associated with elongation of axial length longer than 26 mm or refractive error at least-6 diopter.

High myopia is one of the most prevalent refractive condition globally with a higher risk of other eye conditions Moreover in high myopic eyes the incidence of cataract is significantly higher than in non myopic eyes and the progression is also faster.

Calculation of IOL in high myopic eyes remains a challenge often leading to unexpected postoperative hyperopia the main potential sources of errors in IOL calculation for high myopic eyes include AL measurement & IOL constants used &IOL power calculation formula used.

investigators suspect that the SRK I1 formula is inaccurate for myopic eyes, and that new formulas are needed, taking into account all those factors that make up the dioptric power of an eye.

Formulas for IOL power calculation had past four generations, first generation formulas were theoretical and based on the same fundamental constant with no respect to anterior chamber depth. Since then, Binkhorst, Holladay, Hoffer and Shammas had refined the existing theoretical formulas where each of them developed his regression formula based on analysis of their previous IOL cases .

This work was amalgamated in 1980 and yielded the Sanders Retzlaff Kraff I (SRKI) formula The second generation was designed by combining linear regression analysis and stepwise adjustment for long and short eyes according to anterior chamber depth .

The third and fourth generation formulas, started by Holladay in 1988, all aimed at better calculation of the IOL power in eyes with extreme axial length where another term had appeared which is IOL specific anterior chamber depth .

The accuracy of third and fourth generation formulas for IOL calculation in patients with high axial myopia had not been fully evaluated For that, the need for more studies conducted to evaluate such accuracy is crucial.

This study will be conducted to evaluate the accuracy of different formulas used for IOL power calculation in patients with high axial myopia undergoing cataract surgery

ELIGIBILITY:
Inclusion Criteria:

- 1- patients with clear lense extraction or cataract & high myope with{ AL more than 26 mm.

2-their IOLpower is less than 15 diopter or their refraction before operation is more than -6.

Exclusion Criteria:

1. Keratoconus patients or those with irregular cornea
2. Patients with post operative complications like posterior capsule injury or vitrous loss.
3. patients who had undergone previous intraocular surgery at anterior segment or posterior segment.

Ages: 30 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: data will be collected from all patients who meet inclusion criteria
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
accuracy of iol power in high myopia | one year
  biometry assment of IOLpower

IPD SHARING:
Plan to Share IPD: Undecided
Evaluation of accuracy of IOL power calculation in high myopia.